CLINICAL TRIAL: NCT03821974
Title: The Comparison of Wet Suction Technique and Dry Suction Technique in Endoscopic Ultrasound-guided Fine-needle Aspiration (EUS-FNA) for the Outcomes in Pancreatic Solid Lesions: a Prospective, Randomized Controlled, Blinded Trial
Brief Title: The Comparison of Wet Suction and Dry Suction Technique in EUS-FNA for the Outcomes in Pancreatic Solid Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: EUS2019-001
Record Dates: First submitted 2019-01-15; First posted 2019-01-30 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Pancreatic Solid Lesions
Keywords: Pancreatic solid lesions; wet suction technique; dry suction technique

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dry group (Experimental): The sequence of the technique of the puncture is dry-wet-dry-wet.
  Interventions: Procedure: wet suction technique; Procedure: dry suction technique
- wet group (Experimental): The sequence of the technique of the puncture is wet-dry-wet-dry.
  Interventions: Procedure: wet suction technique; Procedure: dry suction technique

INTERVENTIONS:
Procedure: wet suction technique — For the wet suction technique, after removing the stylet, the needle was flushed with 2 mL of saline solution to replace the column of air with saline solution. A 10-mL suction syringe, loaded to 5ml negative pressure, was attached in a "locked" position to the needle after flushing the needle with saline solution. The needle is moved back and forth 20-30 times by applying negative pressure suction within the lesion. Afterwards, the needle is withdrawn from the lesion.
Procedure: dry suction technique — For the dry suction technique, after locating by EUS, the stylet was removed from the needle before performing FNA. A 10-mL syringe, loaded to 5ml negative pressure, was attached in a "locked" position to the needle. Suction was applied after the lesion was punctured. The needle is moved back and forth 20-30 times by applying negative pressure suction within the lesion. Afterwards, the needle is withdrawn from the lesion.

SUMMARY:
The objective of this randomized controlled trial is to evaluate whether wet suction technique (WST), compared with dry suction technique (DST), shall present a better outcome with regard to the diagnostic yield and specimen quality of patients with solid lesions in the pancreatics.

DETAILED DESCRIPTION:
Endoscopic ultrasound guided fine-needle aspiration (EUS-FNA) has become an inevitable indispensable method for acquiring a pathological diagnosis in a variety of clinical conditions. It has been widely used due to the high sensitivity, specificity and safety. In order to improve the puncture efficiency of FNA, many domestic and oversea scholars have conducted several clinical trials. Among them, there are many studies on the type of needle, needle pattern, slow pull or vacuum suction, and there are only two related reports on wet suction (saline) and dry suction technique. There still have many controversies in the researchers about which technique is more dominant in the wet or dry suction. The wet suction technique is relying on pre-flushing the needle with saline to replace the column of air with fluid followed by aspiration at the proximal end, using a prefilled suction syringe with saline. It has been suggested that the presence of a saline-solution column might keep the needle from getting clogged while avoiding the inherent inconvenience of a metal stylet, so that it can improve the quality of specimens, diminish the contamination of blood, and increase the diagnostic yield and accuracy. Wet suction may become the development trend of EUS-FNA in the future because the application of wet suction is expected to improve the diagnostic efficiency and the quality of samples in FNA.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years, < 80 years
2. female or male
3. Patients are required to undergo EUS-FNA after undergoing imaging examination (MRI, CT, or ultrasonography) which identify that the pancreatic lesions are existing and solid.
4. Agree to attend this study and signed informed consent letter

Exclusion Criteria:

1. bad physical condition, including hemoglobin ≤ 8.0 g/dl, severe cardiorespiratory dysfunction, and so on
2. Coagulopathy (platelet count < 50,000/mm3, international normalized ratio > 1.5) or having taken oral anticoagulation agents such as aspirin or warfarin in the previous week
3. Be rejected by anesthesia
4. Acute pancreatitis in the previous 2 weeks
5. Pregnant or lactation period
6. Psychiatric disease, drug addiction, or other reason for unreliable follow-up or questionnaires
7. Don't agree to attend this study and absence of informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
The primary outcome is defined as the overall diagnosis yield of solid lesions by EUS-FNA with each aspiration technique. | 20 weeks
  The primary outcome is defined as the overall diagnosis yield of solid lesions by EUS-FNA with each aspiration technique.

SECONDARY OUTCOMES:
The second outcome is defined as the diagnose yield of first pass of solid lesions by EUS-FNA with each aspiration technique. | 20 weeks
  The second outcome is defined as the diagnose yield of first pass of solid lesions by EUS-FNA with each aspiration technique.
The third outcome is the diagnose yield in benign solid lesions by EUS-FNA with each aspiration technique. | 20 weeks
  The third outcome is the diagnose yield in benign solid lesions by EUS-FNA with each aspiration technique.
The forth outcome is the diagnose yield in malignant solid lesions by EUS-FNA with each aspiration technique. | 20 weeks
  The forth outcome is the diagnose yield in malignant solid lesions by EUS-FNA with each aspiration technique.
The fifth outcome is the diagnose yield in solid lesions in different parts of the pancreas by EUS-FNA with each aspiration technique. | 20 weeks
  The fifth outcome is the diagnose yield in solid lesions in different parts of the pancreas by EUS-FNA with each aspiration technique.

CONTACTS AND LOCATIONS:
Overall Officials: Li Tian, MD, Principal Investigator — The Third Xiangya Hospital of Central South University; Ting Tong, MD, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- The third Xiangya Hospital of central south University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No